CLINICAL TRIAL: NCT00877149
Title: A Single-arm, Multicenter, Open-label, 52-week Treatment, Extension Study to CLDT600ACN04 Study to Evaluate the Efficacy (Including Histological Improvement) and Safety in Fourth to Sixth Year of Telbivudine Treatment in Patients With Chronic Hepatitis B
Brief Title: Efficacy of Telbivudine Treatment at Long Term on the Absence of Liver Inflammation in Patients With Compensated Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600ACN04E1
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Compensated Chronic Hepatitis B
Keywords: Chronic HBV
MeSH Terms: interventions — Telbivudine

ARMS (1):
- A (Experimental)
  Interventions: Drug: telbivudine/LDT600

INTERVENTIONS:
Drug: telbivudine/LDT600

SUMMARY:
The purpose of this trial is to provide data of absence of inflammation in patient liver histology after long-term telbivudine treatment and thus help investigators to make a comprehensive judgment on treatment discontinuation in selected patients

ELIGIBILITY:
Inclusion Criteria:

* Patient completed study CLDT600ACN04 study and will be available to immediately rollover into this study without discontinuation of study drug.
* Patient was not discontinued from the previous CLDT600ACN04 study.
* Adult patients with CHB (HBeAg positive or HBeAg negative).
* HBV DNA PCR undetectable in recent 12 months.

Exclusion Criteria:

* Pregnant or breastfeeding, or has plan of pregnant during study period.
* Patient is co-infected with hepatitis C virus (HCV), hepatitis D virus (HDV), or HIV at screening visit.
* Patient has received within the past 12 months any anti-HBV treatment combination (add-on therapy) or switch to other anti HBV treatment from Telbivudine at investigator's discretion.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess proportion of patients with absence of inflammation in liver biopsy at study entry and combine the histological assessment with serological evaluations. | Visit 2 (week 1)

SECONDARY OUTCOMES:
To assess the HBV DNA PCR negativity at 4th-6th year treatment with telbivudine (LDT), in selected patients who have completed study CLDT600ACN04 and will continue telbivudine treatment | weeks 1, 24, 52 and 24 weeks post-treatment
To evaluate the percentage of patients with HBeAg loss and/or gain of detectable level of HBeAb in HBeAg positive CHB at baseline of NV-02B-007 or NV-02B-015 studies | weeks 24 and 52, 24 weeks post-treatment
To evaluate percentage of patients with with HBsAg loss and/or HBsAg seroconversion | weeks 24, 52 and 24 weeks post-treatment
To evaluate the changes in Knodell inflammatory and fibrosis scores from biopsy at study entry compared to biopsy at baseline of studies NV-02B-007 and NV-02B-015 | Visit 2 (week 1)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- China (4):
  - Beijing Ditan Hospital, Beijing
  - First Hospital of Peking University, Beijing
  - Peking University People's Hospital, Beijing
  - Ruijin Hospital, Affiliated to 2nd Medical university, Shanghai

REFERENCES:
- [Derived] Hou JL, Xu D, Shi G, Wan M, Goodman Z, Tan D, Xie Q, Chen C, Wei L, Niu J, Wang Q, Ren H, Wang Y, Jia J, Bao W, Dong Y, Trylesinski A, Naoumov NV. Long-Term Telbivudine Treatment Results in Resolution of Liver Inflammation and Fibrosis in Patients with Chronic Hepatitis B. Adv Ther. 2015 Aug;32(8):727-41. doi: 10.1007/s12325-015-0232-2. Epub 2015 Sep 2. PMID 26329749